CLINICAL TRIAL: NCT02049008
Title: Clinical, Microbiological and Immunological Effects of Antimicrobial Photodynamic Therapy on Non-surgical Treatment of Aggressive Periodontitis: a Double-blind Split-mouth Randomized Controlled Clinical Trial.
Brief Title: Treatment of Aggressive Periodontitis With Repeated Adjunctive Antimicrobial Photodynamic Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Michel Reis Messora, Ph.D., University of Sao Paulo
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012/13260-8 FAPESP
Record Dates: First submitted 2013-12-09; First posted 2014-01-29 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Aggressive Periodontitis
MeSH Terms: conditions — Aggressive Periodontitis | interventions — Photochemotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Photodynamic Therapy (Experimental)
  Interventions: Other: Photodynamic Therapy
- Sham Photodynamic Therapy (Sham Comparator)
  Interventions: Other: Sham Photodynamic Therapy

INTERVENTIONS:
Other: Photodynamic Therapy — After a full-mouth scaling and root planning (SRP), the periodontal pockets of teeth selected to receive antimicrobial photodynamic therapy (aPDT) will be irrigated with distilled water. Shortly thereafter, the dye will be applied (phenothiazine hydrochloride- 10mg/mL) from the bottom of the pocket. After 1 minute, irrigation will be performed with distilled water to remove the excess of dye. The stained area will be irradiated with a diode laser (660 nm and a 60 mW/cm²). Six sites per tooth under treatment will be irradiated (10 seconds/ site). The applications of aPDT will be repeated in the same way until the second week (days: 2, 7,14). Before the application, the supragingival plaque will be removed.
  Arms: Photodynamic Therapy
Other: Sham Photodynamic Therapy — After a full-mouth scaling and root planning (SRP), the periodontal pockets of teeth selected will receive a simulation of antimicrobial photodynamic therapy (aPDT): irrigation with distilled water and simulated laser application. The simulations of aPDT will be repeated in the same way until the second week (days: 2, 7,14). Before the application, the supragingival plaque will be removed.
  Arms: Sham Photodynamic Therapy

SUMMARY:
The treatment of aggressive periodontitis (AgP) represents a challenge for clinicians, because there are no standardized protocols for efficient control of the disease. The aim of this study is to evaluate the effect of multiple applications of antimicrobial photodynamic therapy (aPDT) as an adjunct to non-surgical periodontal treatment (nsPT) in patients diagnosed with AgP. Twenty patients with a clinical diagnosis of AgP will be treated in a split-mouth design study to either aPDT associated with scaling and root planning (SRP) or SRP only. aPDT will be performed by using a laser light source with 690 nm wavelength associated with a phenothiazine photosensitizer. The applications will occur in four episodes (days 0, 2, 7 and 14). All patients will be monitored for 90 days. Clinical assessment of plaque index, probing depth, clinical attachment level and bleeding on probing will be performed at baseline (pre-intervention period) and 30 and 90 days after the nsPT. Subgingival plaque samples will be collected (at baseline and 30 and 90 days after the nsPT) and the counts of 40 subgingival species will be determined using DNA-DNA checkerboard hybridization. Gingival crevicular fluid samples will be collected (at baseline and 14, 30 and 90 after the nsTP) for evaluation the volume of fluid (Periotron) and the levels of Interleukin 1 beta, Interleukin 10 and Tumor Necrosis Factor alpha (Luminex). Data obtained will be statistically analyzed.

DETAILED DESCRIPTION:
Non-Surgical Periodontal Therapy

Seven days prior to the non-surgical periodontal therapy, periapical radiographs will be taken from the whole mouth of all patients. They will be set in an oral hygiene program (OHP) according to their specific needs. In this program, patients will be instructed about an effective self-performed plaque control, including information about the Bass Technique (Bass, 1954) and interproximal cleaning with dental floss and interdental brushes. They will be also motivated to brush the dorsal surface of the tongue once a day and will receive a dentifrice that shall be used throughout the experimental period (Colgate Total®, Anakol Ind. Com Ltda - Brazil's Kolynos - Colgate Palmolive Co., Sao Bernardo do Campo, SP, Brazil). After the OHP, subjects will undergo the assessment of clinical periodontal parameters previously described and the collection of subgingival plaque and GCF in selected sites (baseline) will be performed. Shortly, patients will receive supragingival scaling and coronal polishing with prophy cup on all the teeth present in the oral cavity. The non-surgical periodontal therapy will initiate 7 days after the OHP and initial supragingival scaling. Within 24 hours, a specialist in Periodontics will perform supra and subgingival scaling and root planing of all teeth with periodontal involvement, using hand (Gracey Curettes, Hu-Friedy, Chicago, IL, USA) and ultrasonic instruments. The instrumentation will be performed on each quadrant until achievement of an adequate cleaning and root planing, which will be verified with a dental explorer. Individuals will receive professional prophylaxis biweekly during three months after the end of the nonsurgical periodontal therapy. On biweekly follow-up visits, patient's cooperation will be monitored by verifying the status of oral hygiene.

Antimicrobial photodynamic Therapy

After a full-mouth scaling and root planning (SRP), the periodontal pockets of teeth selected to receive antimicrobial photodynamic therapy (aPDT) will be irrigated with distilled water. Shortly thereafter, the dye will be applied (phenothiazine hydrochloride- 10mg/mL) from the bottom of the pocket. After 1 minute, irrigation will be performed with distilled water to remove the excess of dye. The stained area will be irradiated with a diode laser (660 nm and a 60 mW/cm²). Six sites per tooth under treatment will be irradiated (10 seconds/ site). The applications of aPDT will be repeated in the same way until the second week (days: 2, 7,14). Before the application, the supragingival plaque will be removed.

Each patient will be impressed with alginate in order to obtain models of the dental arches and elaborate a guide plate made of acetate. This plate will present grooves that will be used as references to standardize the insertion and tilt of the automated periodontal probe (Florida Probe System, Florida Probe Corporation, Gainesville, FL, USA). The visible plaque index for each patient, rated dichotomously (O'Leary et al. 1972), will be determined by the percentage of tooth surfaces with deposits of plaque stained with disclosing solution.

Clinical monitoring

The following clinical periodontal parameters will be assessed at 6 sites of each tooth (mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual and disto-lingual): (i) probing pocket depth (PPD): it will be measured from the gingival margin to the bottom of the pocket; (ii) gingival recession (GR): it will be measured from the enamelcement junction to the bottom of the pocket; (iii) clinical attachment level (CAL): it will be measured as PPD + GR (GR will be equal to 0 whenever the cementenamel junction is covered); (iv) bleeding on probing (BOP): it will be evaluated dichotomously: the presence of the bleeding will be considered positive when occurring within 30 seconds from the insertion of the probe for probing depth; (v) Plaque index (PI): it will be evaluated dichotomously. BOP, PPD, CAL and GR will be measured at six sites per tooth (mesio-buccal, buccal, disto-buccal, disto-lingual, lingual and mesio-lingual). All probing measurements will be performed using an automated periodontal probe.

The clinical periodontal parameters and the plaque index of each patient will be recorded at baseline (pre-intervention), as well as +30 and +90 days after the non-surgical periodontal therapy. The Kappa index will be used to evaluate the examiner calibration on clinical periodontal parameters collection in order to calculate the intra-examiner agreement. According to the World Health Organization (WHO) criteria for diagnosis, the acceptable Kappa index of agreement must be greater than or equal to 0.85 (WHO, 1997). This level of agreement will be used for calibration of the examiner in this project. Ten patients, each one showing at least two pairs of contralateral single-rooted teeth with PD ≥ 5 mm on interproximal sites, will be selected to calibrate the examiner. Each patient will be evaluated on two separate occasions 48 hours apart in order to obtain the intra-examiner reliability through the Kappa index.

Immunological monitoring

At baseline and +14 and +30 and +90 days after the non-surgical periodontal therapy, GCF samples will be obtained from eight interproximal sites of each patient. The supragingival plaque from selected teeth will be removed and the sites will be carefully dried with air jets, and subsequently isolated with sterile cotton rolls. Samples of GCF will be obtained with papers strips (Periopaper® -Oralflow Inc., Amityville, NY, USA). The papers strips will be gently inserted into the orifice of the periodontal pocket, remaining 30 seconds subgingivally. The amount of GCF absorbed will be determined by an electronic measurer of humid mass (Periotron® -Oralflow Inc., Amityville, NY, USA). Samples will be placed in sterile Eppendorf tubes stored at - 80°C for cytokines (IL-1β, IL-10 and TNF-a) quantification (pg/μl) at Genese Laboratory (Genese Produtos Diagnosticos LTDA, Sao Paulo, SP, Brazil). Cytokines levels will be determined using a three-plex Millipore kit (Millipore Corporation, Billerica, MA, USA) and the Luminex 100TM system (Luminex, MiraiBio, Alameda, CA, USA).

Microbiological monitoring

At baseline and +30 and +90 days after the non-surgical periodontal therapy, samples of subgingival plaque will be obtained from eight interproximal sites of each patient. Samples will be individually analyzed for their content of 40 subgingival bacterial species using the checkerboard DNA-DNA hybridization technique (Socransky et al., 2004a; Socransky et al., 2004b). The selected teeth will be isolated with sterile cotton rolls and dried with air jets. Then, the supragingival plaque will be carefully removed using a sterile curette. Another sterile curette will be used to collect the subgingival plaque, starting from the bottom of the periodontal pocket to its coronal portion. The samples will be stored in sterilized Eppendorf tubes and will be processed at the Microbiology Laboratory of the Guarulhos University (UNG, Guarulhos, SP, Brazil).

Statistical analysis

The normality and homoscedasticity of the data obtained will be checked. Comparisons within groups and among groups at different time intervals will be performed through parametric or non-parametric appropriate tests. The significance level will be set at 5% in all tests. All calculations will be performed by SPSS software (SPSS, Chicago IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* subjects with <35 years old;
* a minimum of 20 teeth present;
* two pairs of single-rooted teeth in opposite sides with proximal sites showing probing depth and clinical attachment level ≥ 5 mm.

Exclusion Criteria:

* Positive history of antibiotic-therapy in the last six months;
* Positive history of basic periodontal treatment in the last six months;
* Systemic disease that can interfere with the progression of disease or response to treatment (eg, diabetes, immune disorders);
* Extensive prosthetic involvement;
* Need for antibiotic prophylaxis for performing routine dental procedures;
* Use of anti-inflammatory drugs for long periods of time;
* Smoking
* Pregnancy.

Max Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in clinical attachment level at +90 days. | The clinical periodontal parameter will be recorded at baseline (pre-intervention) and +90 days after the non-surgical periodontal therapy.

SECONDARY OUTCOMES:
Change from baseline in counts of 40 subgingival bacterial species at +30 and +90 days | Microbiological monitoring (at baseline and +30 and +90 days after the non-surgical periodontal therapy) using the checkerboard DNA-DNA hybridization
Change from baseline in levels of IL-1β, IL-10 and TNF-alpha at +14 and +30 and +90 days | Immunological monitoring (at baseline, +14 and +30 and +90 days after the non-surgical periodontal therapy) using Luminex.
Numbers of patients requiring additional periodontal treatment at +90 days. | Considering each group separately, it will be evaluate the number of patients presenting at least a site with PPD≥5 mm and positiveBOP at 90 days post-therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Michel R Messora, Dr., Principal Investigator — University of São Paulo - Ribeirão Preto
Locations (1):
- School of Dentistry of Ribeirao Preto - University of São Paulo, Ribeirão Preto, São Paulo, Brazil